CLINICAL TRIAL: NCT06028724
Title: A Prospective, Observational Study on the Prevalence of Clinically Useful Mutations in Solid Tumor Characterized by Next Generation Sequencing Methods on Liquid Biopsy Analysis (POPCORN)
Brief Title: A Study on the Prevalence of Clinically Useful Mutations in Solid Tumor Characterized by Next Generation Sequencing Methods on Liquid Biopsy Analysis (POPCORN)
Acronym: POPCORN
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2022-51
Record Dates: First submitted 2023-08-03; First posted 2023-09-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor; Advanced Solid Tumor; Locally Advanced Solid Tumor; Colon Rectal Cancer; Gastric Cancer; Pancreatic Cancer; Bile Duct Cancer; Hepatocarcinoma; Breast Cancer; Ovarian Cancer; Endometrial Cancer; Cervical Cancer; Vulva Cancer; Melanoma
MeSH Terms: conditions — Colonic Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Bile Duct Neoplasms; Carcinoma, Hepatocellular; Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The implementation of liquid biopsy in clinical practice has been favored by the rapid development of genome sequencing techniques designed to analyze mutations in ctDNA. Among these, the Next generation sequencing (NGS) is a technique that consists in sequencing several genomes in a short time span, collecting information about a wider range of genomic alterations, using small quantities of genetic material. It is used to identify potential circulating dynamic biomarkers of treatment sensitivity or resistance in a real word multi-pathology evaluation. In this way, defining the mutational status of clinical relevance genes in real world, as a predictive biomarker to identify those patients most likely to benefit from target therapy, offers the potential to optimize access to further therapies. The aim of this study is to evaluate the real-world prevalence of clinically useful mutations in patients who are receiving therapy for advanced and locally advanced solid tumor through liquid biopsy.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

* Patients, 18 years of age or older
* Competent and able to comprehend, sign and date an Ethics Committee (EC) approved Informed Consent Form (ICF) before performance of any study-specific procedures or tests
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Histologically proven diagnosis solid tumor
* Diagnosis of advanced or locally advanced disease
* Patients candidated to receive standard therapy in the following line:
* first, second or third-line therapy for colon-rectal cancer in IV stage
* first or second-line therapy for gastric cancer in IV stage
* primary intent or first-line therapy for pancreatic cancer
* first-line therapy for bile duct cancer
* first or second-line therapy for hepatocarcinoma
* first, second, third, fourth or fifth-line therapy for breast cancer in IV stage
* chemotherapy for ovarian cancer in advanced stage (FIGO III-IV) and at the time of first relapse
* first or second-line therapy for endometrial cancer in advanced stage (FIGO III-IV)
* first or second-line therapy for advanced or locally advanced cervical cancer
* therapy for locally advanced or first line therapy for metastatic vulva cancer
* first, second or third-line therapy for melanoma (third-line therapy only in BRAF-mutated melanoma)

Exclusion Criteria:

* Diagnosis of any secondary malignancy within the last 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* Patients unable or unwilling to undergo as per protocol assessments at the four planned timepoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are receiving therapy for advanced and locally advanced solid tumor as specified in eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 782 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Real world prevalence of clinically useful mutations in solid tumors | at the beginning of treatment
  Real world prevalence of clinically useful mutations in solid tumors, defined as the proportion of patients with the detection of clinically useful mutations through ctDNA NGS, at the beginning of systemic therapies defined as per inclusion criteria for advanced disease.

SECONDARY OUTCOMES:
To identify emerging gene alterations associated with Progression Free Survival | from study enrollment until progression or death for any cause, up to 7 years
  To identify emerging gene alterations associated with Progression Free Survival (PFS) defined as the time from study enrollment until progression or death for any cause, whichever comes first
To identify emerging gene alterations associated with Overall Survival | from study enrollment until death for any cause, up to 7 years
  To identify emerging gene alterations associated with Overall Survival, defined as the time from study enrollment until death for any cause
To describe changes in ctDNA associated biomarkers during treatment | up to 7 years
  Difference in frequency of patients with ctDNA associated biomarkers at different time point during treatment (at baseline, at start of cycle 2, at first radiological evaluation, at relapse or end of follow-up)
To evaluate the association between somatic genetic alterations and the histopathological features of the tumor | up to 7 years
  Frequency of somatic genetic alterations in subgroups of patients with different histopathological tumor characteristics
To evaluate the association between somatic genetic alterations and pattern of metastasis | up to 7 years
  Frequency of somatic genetic alterations in subgroups of patients with metastasis
To evaluate the association between somatic genetic alterations and the clinical characteristic of the enrolled patients | up to 7 years
  Frequency of somatic genetic alterations in subgroups of patients with different clinical characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Puglisi, MD, PhD, Principal Investigator — IRCCS-Centro di Riferimento Oncologico (CRO), Aviano (PN)
Locations (1):
- IRCCS, Centro di Riferimento Oncologico (CRO) di Aviano, Aviano, Pordonone, Italy